CLINICAL TRIAL: NCT01102985
Title: An Exercise Intervention to Improve Health in Postmenopausal Cancer Survivors
Brief Title: Women With Cancer: An Exercise Study to Promote Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0801003383; 1R01CA122658-01A2 (NIH)
Record Dates: First submitted 2010-01-19; First posted 2010-04-13 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Bone Loss; Cancer
Keywords: exercise; physical activity; intervention; cancer survivor
MeSH Terms: conditions — Bone Diseases, Metabolic; Neoplasms; Motor Activity | interventions — Exercise; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic resistance (Experimental): 12 month aerobic resistance exercise at a fitness center
  Interventions: Behavioral: aerobic resistance exercise
- home based physical activity (Active Comparator): national recommendations for physical activity for adults
  Interventions: Behavioral: home based health promotion

INTERVENTIONS:
Behavioral: aerobic resistance exercise — three times per week aerobic resistance exercise for 12 months
  Other Names: physical activity
  Arms: aerobic resistance
Behavioral: home based health promotion — education and support to adapt national guidelines for 30 minutes physical activity most days of the week
  Other Names: health promotion
  Arms: home based physical activity

SUMMARY:
The purpose of the study is to evaluate the effect of an aerobic-resistance exercise program compared to a home based physical activity program on bone mass, body composition, metabolic risk factors and cardiovascular fitness in women with cancer who have completed therapy.

DETAILED DESCRIPTION:
The proposed study will evaluate an endurance-resistive exercise intervention to attenuate the effects of menopause and cancer treatment (bone loss, increased body fat, decreased lean muscle mass, weight gain, decreased physical activity) in an at-risk population of female cancer survivors. Women with solid tumors (breast, gynecological, colo-rectal) and lymphoma who have completed primary and/or adjuvant therapy within the past three years and who are perimenopausal or early postmenopausal and any woman on an Aromatase Inhibitor will be recruited to participate in a randomized controlled trial (RCT) of a 12 month exercise intervention (N=75) versus a health promotion control group (N=75). The specific aims of the study are to: (1) examine the effects of an exercise intervention on bone mass (serum biomarkers, lumbar spine, hip DEXA) and body composition (whole body DEXA, weight, waist circumference), (2) examine the effect of an exercise intervention on metabolic risk factors (lipids, cholesterol, fasting glucose, insulin resistance, Hemoglobin A1-C, and blood pressure), and (3) examine the effects of an exercise intervention on functional status and cardiovascular fitness (exercise stress test).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Cancer diagnosis
* Postmenopausal

Exclusion Criteria:

* Health condition contraindication to moderate physical activity

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Bone mass-lumbar spine and hip (DEXA) | baseline, 12 months
  Serum biomarkers for bone (serum NTX and serum osteocalcin) will be drawn at baseline, 6 and 12 months. Bone mass for lumbar spine and hip will be measured by DEXA scan at baseline and 12 months.

SECONDARY OUTCOMES:
body composition-% fat mass, % lean muscle mass (whole body DEXA) | baseline, 6, 12 months
  Body composition will be assessed by waist circumference and whole body DEXA scan (% fat mass, % lean muscle mass) at baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Tish Knobf, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Knobf MT, Jeon S, Smith B, Harris L, Thompson S, Stacy MR, Insogna K, Sinusas AJ. The Yale Fitness Intervention Trial in female cancer survivors: Cardiovascular and physiological outcomes. Heart Lung. 2017 Sep-Oct;46(5):375-381. doi: 10.1016/j.hrtlng.2017.06.001. Epub 2017 Aug 10. PMID 28803675